CLINICAL TRIAL: NCT01186731
Title: A Multicenter, Open-Label, Phase II Study of LE-DT for Efficacy and Safety in Patients With Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Efficacy and Safety Study of LE-DT to Treat Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Protocol LE-DT 202
Record Dates: First submitted 2010-08-18; First posted 2010-08-23 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-08

CONDITIONS: Pancreatic Cancer
Keywords: SPARC (secreted protein acid rich in cysteine); serum Carbohydrate Antigen CA 19-9
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liposome Entrapped Docetaxel (LE-DT) (Experimental)
  Interventions: Drug: Liposome Entrapped Docetaxel (LE-DT)

INTERVENTIONS:
Drug: Liposome Entrapped Docetaxel (LE-DT) — 110 mg/m2 (IV)in vein on day 1 of each 21 day cycle , 6 cycles, until progression or unacceptable toxicity
  Other Names: Liposomal Docetaxel; LE-DT

SUMMARY:
LE-DT is a novel, proprietary delivery system of docetaxel developed by NeoPharm, Inc. Docetaxel (currently marketed as Taxotere) is an anti-microtubule agent that prevents cell division. By removing toxic detergent used in Taxotere, the form of LE-DT, shows reduced toxicity and comparable therapeutic efficacy in pre-clinical study. The clinical evidence obtained from the NeoPharm Phase I study shows fewer side effects and possibly administered at higher dose to induce greater effectiveness of LE-DT. In addition, docetaxel has shown positive activity of protein bound taxane therapy in treating patients with pancreatic cancer. The current Phase II study is designed to accomplish the following objectives:

1. Assess the antitumor effect of 110 mg/m2 LE-DT administered intravenous (IV) every three weeks in pancreatic cancer patients with locally advanced or metastatic disease
2. To evaluate the progression-free survival and overall survival
3. To correlate secreted protein acid rich in cysteine expression with tumor response
4. To evaluate the safety of LE-DT, in particular peripheral neuropathy, water retention as well as myelotoxicity
5. To correlate pharmacogenetic variations in patients with LE-DT pharmacodynamic endpoints, including toxicities.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years or older, male and female.
2. Patient has histopathologically confirmed diagnosis of adenocarcinoma of the pancreas. Patients with islet cell neoplasms are excluded. Biopsy sample must be available for SPARC assay.
3. Patients must have clinical or radiographic evidence of locally advanced or metastatic pancreatic cancer with measurable disease.
4. Male or non-pregnant and non-lactating female:

   * If a female patient is of child-bearing potential, as evidenced by regular menstrual periods, she must have a negative serum pregnancy test (β hCG) documented within 72 hours of the first administration of study drug.
   * If sexually active, the patient must agree to use contraception considered adequate and appropriate by the Investigator.
5. Patient can be newly-diagnosed without prior treatment or have failed initial adjuvant treatment with either gemcitabine, 5-FU or capecitabine with or without radiation therapy.
6. Patient has the following blood counts at baseline:

   * ANC greater than or equal to 1500 per uL
   * Platelets greater than or equal to 100000 per uL
   * Hgb greater than or equal to 9 g per dL
7. Patient has the following blood chemistry levels at baseline:

   * AST (SGOT), ALT (SGPT) less than or equal to 2.5 times of the upper limit of normal range (ULN), unless liver metastases are present, then less than or equal 5 times of the ULN is allowed
   * Bilirubin less than or equal to 1.5 times of the ULN
   * Serum creatinine less than or equal to 1.5 times of the ULN or calculated clearance greater than or equal to 60 mL/min for patients with serum creatinine levels above the institutional normal value.
8. Patient has acceptable coagulation profile as indicated by a Prothrombin time (PT) and Partial Thromboplastin Time (PTT) within normal limits (plus or minus 15%) unless explained by the use of anticoagulants
9. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status 0-2
10. Patient has one or more metastatic lesions or locally advanced primary tumor measurable by CT or MRI.
11. Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board-approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

1. Patient has known brain metastases.
2. Patient has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
3. Patient has known infection with HIV, hepatitis B, or hepatitis C.
4. Patient has undergone major surgery, other than diagnostic surgery (i.e. surgery done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to Day 1 of treatment in this study.
5. Patient who have received any other treatment for pancreatic cancer including radiotherapy, chemotherapy or any investigational therapy with the exception of initial adjuvant treatment including either gemcitabine, 5-FU or capecitabine with or without radiation therapy
6. Patient has a history of allergy or hypersensitivity to the study drug.
7. Patient has serious medical risk factors involving any of the major organ systems such that the Investigator considers it unsafe for the patient to receive an experimental research drug.
8. Patient has pre-existing peripheral neuropathy of Grade >1 based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
9. Patient is unwilling or unable to comply with study procedures.
10. Patient is enrolled in any other clinical or investigational trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Response rate of tumor size reduction at 110 mg/m2 LE-DT dose level | 1 year
  Measurable disease response will be assessed by radiographic method, CT or MRI, along with serum CA 19-9 after completed 2, 4 and 6 cycle.

SECONDARY OUTCOMES:
SPARC tumor expression following the treatment of LE-DT at 110 mg/m2 dose level | 1 year
  SPARC tumor expression will be assessed as a potential predictor of tumor response

CONTACTS AND LOCATIONS:
Overall Officials: John L Marshall, M.D., Principal Investigator — Lombardi Cancer Center, Georgetown University Medical center
Locations (1):
- Lombardi Cancer Center, Georgetown University Medical Center, Washington D.C., District of Columbia, United States